CLINICAL TRIAL: NCT07354412
Title: Investigating Cannabis Use Parameters on Anesthesia and Inflammation in Lumbar Spinal Surgeries
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Pias Malaker, Principal Investigator, University of Missouri-Columbia
Other Study IDs: 2128606
Record Dates: First submitted 2025-06-09; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use
Keywords: cannabis; anesthesia; inflammation; cytokines
MeSH Terms: conditions — Marijuana Abuse; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Never users: Patients who have never used cannabis products
- Current users: Individuals who have used cannabis products in the last 30 days
- Past users: Individuals who have used cannabis products in the past but not in the last 30 days

SUMMARY:
Cannabis is the most commonly used illicit drug in the United States with reported rates of use increasing from approximately 50 million in 2020 to 61.8 million in 2023 among individuals aged 12 or older. This rise can be attributed to a combination of growing social acceptance and expanding legalization for recreational and medical use of cannabis. Consequently, this has led to increased commercially available cannabis products with heterogeneous concentrations of cannabinoids (i.e., THC:CBD ratios) and new methods of administration becoming more available (e.g., vaping and gummies). Taken together, this rapidly shifting landscape further contributes to the significant variability in individual use patterns (i.e., frequency, duration, and route of administration) resulting in diverse clinical responses, which poses significant challenges for anesthetic management. Recent systematic reviews and meta-analysis have quantitatively demonstrated that cannabis users require higher dosages during anesthesia induction, experience greater hemodynamic instability, and report higher opioid consumption and pain scores post-operatively. These findings have led to the prevailing notion that cannabis exposure adversely affect anesthetic management. Yet, key cannabis exposure parameters in individual use patterns (i.e., variations in THC:CBD ratios, route of administration, frequency, and duration of use) remain poorly characterized and could confound observed clinical effects in relation to their effects on pain modulation and anesthetic requirements. Current perioperative assessments do not account for these critical variables, creating a gap that limits the development of more accurate and personalized anesthetic protocols. Failure to account for individual cannabis exposure parameters may lead to inappropriate anesthetic dosing - where underdosing could result in intraoperative awareness, pain, or patient movement, while overdosing might cause cardiovascular depression, respiratory failure, or prolonged recovery from anesthesia. Concomitantly, researchers have discovered that cannabis consumption modulates immune function such that early life exposure to cannabis produces a long-lasting and persistent inflammatory state characterized by reduced serum levels of IL-6, TNF-α, and IL-2. In contrast, recent research demonstrates that cannabinoid exposure improves skin healing in patients with cutaneous disorders. However, the effects of altered inflammatory responses, and the diverse actions of various cannabinoids on postoperative wound healing remain largely unexplored. Our long-term goal is to elucidate the mechanistic impact of chronic cannabis use parameters on anesthetic and analgesic requirements, thereby enabling the development of personalized, evidence-based perioperative management strategies. The investigators hypothesize that chronic cannabis exposure leads to impaired endogenous pain and immune modulation, resulting in increased intraoperative anesthetic dosing, heightened hemodynamic variability, and elevated postoperative pain and inflammation.

DETAILED DESCRIPTION:
Cannabis is the most commonly used illicit drug in the United States with reported rates of use increasing from approximately 50 million in 2020 to 61.8 million in 2023 among individuals aged 12 or older. This rise can be attributed to a combination of growing social acceptance and expanding legalization for recreational and medical use of cannabis. Consequently, this has led to increased commercially available cannabis products with heterogeneous concentrations of cannabinoids (i.e., THC:CBD ratios) and new methods of administration becoming more available (e.g., vaping and gummies). Taken together, this rapidly shifting landscape further contributes to the significant variability in individual use patterns (i.e., frequency, duration, and route of administration) resulting in diverse clinical responses, which poses significant challenges for anesthetic management. Recent systematic reviews and meta-analysis have quantitatively demonstrated that cannabis users require higher dosages during anesthesia induction, experience greater hemodynamic instability, and report higher opioid consumption and pain scores post-operatively. These findings have led to the prevailing notion that cannabis exposure adversely affect anesthetic management. Yet, key cannabis exposure parameters in individual use patterns (i.e., variations in THC:CBD ratios, route of administration, frequency, and duration of use) remain poorly characterized and could confound observed clinical effects in relation to their effects on pain modulation and anesthetic requirements. Current perioperative assessments do not account for these critical variables, creating a gap that limits the development of more accurate and personalized anesthetic protocols. Failure to account for individual cannabis exposure parameters may lead to inappropriate anesthetic dosing - where underdosing could result in intraoperative awareness, pain, or patient movement, while overdosing might cause cardiovascular depression, respiratory failure, or prolonged recovery from anesthesia. Concomitantly, researchers have discovered that cannabis consumption modulates immune function such that early life exposure to cannabis produces a long-lasting and persistent inflammatory state characterized by reduced serum levels of IL-6, TNF-α, and IL-2. In contrast, recent research demonstrates that cannabinoid exposure improves skin healing in patients with cutaneous disorders. However, the effects of altered inflammatory responses, and the diverse actions of various cannabinoids on postoperative wound healing remain largely unexplored. Our long-term goal is to elucidate the mechanistic impact of chronic cannabis use parameters on anesthetic and analgesic requirements, thereby enabling the development of personalized, evidence-based perioperative management strategies. The investigators hypothesize that chronic cannabis exposure leads to impaired endogenous pain and immune modulation, resulting in increased intraoperative anesthetic dosing, heightened hemodynamic variability, and elevated postoperative pain and inflammation. To test this hypothesis, the investigators propose the following specific aims: Specific aim 1: Assess cannabis use parameters of individual use patterns in relation to anesthetic and analgesic requirements during elective spine surgeries. The investigators will conduct a prospective study in patients undergoing ambulatory or short-stay lumbar spine surgery asking them to fill out a survey detailing their individual cannabis use patterns (e.g., frequency, duration, and method of use) and attach pictures of their products (to obtain variations in THC:CBD ratios and product type). The investigators will compare intraoperative anesthetic dosing (e.g., propofol and opioid anesthetics) and evaluate hemodynamic parameters (e.g., blood pressure fluctuations and vasopressor requirements), and assess postoperative pain intensity and analgesic needs between cannabis users and non-users. This aim will provide direct clinical evidence linking specific chronic cannabis exposure parameters to intraoperative anesthetic and analgesic requirements, thereby laying the groundwork for tailored anesthetic protocols to reduce complications during surgery. Specific aim 2: Determine the inflammatory mechanisms by which chronic cannabis use alters pain processing and wound repair. The investigators will measure serum biomarkers of inflammation, including IL-6, TNF-α, IL-2, and CRP before and after surgery, and again at 2- and 6-week follow-up, to assess how chronic cannabis exposure modulates immune responses and wound healing in elective spine surgeries. In parallel, the investigators will obtain subjective pain assessments using validated scales and correlate these with intraoperative anesthetic dosing and inflammatory biomarker levels, thereby elucidating the interplay between cannabis-induced immune modulation in altering pain processing and wound healing. Impact: If successful, these studies will fill critical gaps in our understanding by: • Precisely characterizing how individual cannabis exposure parameters affect perioperative anesthetic and analgesic needs, thereby enabling personalized dosing protocols that reduce the risk of intraoperative awareness, cardiovascular instability, and prolonged recovery. • Defining the immunologic alterations associated with chronic cannabis use and their relationship to wound healing and postoperative pain, which may pave the way for novel interventions to optimize surgical outcomes. This integrative approach will advance the fields of anesthesiology, and surgical perioperative patient care and addiction research.

ELIGIBILITY:
Inclusion Criteria for both cannabis users and non-users:

* Undergoing ambulatory or short-stay lumbar spine surgery.
* English speaking.
* Ability to consent for themselves.
* Aged 18 years and above.
* Access to a smartphone or computer/laptop (to be determined on the day of consent).

Inclusion criteria for cannabis users:

• Any lifetime use of cannabis products irrespective of the strain, CBD/THC content, or frequency of use.

Exclusion Criteria:

* Non-English speaking.
* Inability to consent for themselves.
* Actively pregnant (SOC) or planning to become pregnant in the next 2 months (research only). Urine testing will be done as SOC prior to undergoing surgery.
* Active or past severe psychiatric instability (e.g., active psychosis, acute suicidality)
* Active, uncontrolled use of illicit drugs use such as methamphetamine, cocaine, opioids, etc., as listed in their clinical charts.
* History of major neurological illnesses.
* Presence of an untreated illness or serious medical condition.
* Any other concern that in the investigator's opinion would impact participant safety, study instruction compliance, or confound the interpretation of the study results.
* No access to a smartphone or computer/laptop.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulatory and short-stay lumbar spine surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Propofol dose (mg/kg/hr) | Duration of surgery
  Our primary outcome is intraoperative anesthetic dose (i.e., propofol mg/kg/hr), which will be extracted from anesthesia records and entered into each patient's individual REDCap record by the study personnel.
Change in serum inflammatory biomarker IL-2 (pg/mL) | From enrollment to 6 week post-surgery
  The investigators will measure serum biomarker of inflammation IL-2 (pg/mL) before and after surgery, and again at 2- and 6-week follow-ups, to assess how cannabis exposure modulates immune responses.
Change in serum inflammatory biomarker IL-6 (pg/mL) | From enrollment to 6 week post-surgery
  The investigators will measure serum biomarker of inflammation IL-6 (pg/mL) before and after surgery, and again at 2- and 6-week follow-ups, to assess how cannabis exposure modulates immune responses.
Change in serum inflammatory biomarker TNF-α (pg/mL) | From enrollment to 6 week post-surgery
  The investigators will measure serum biomarker of inflammation TNF-α (pg/mL) before and after surgery, and again at 2- and 6-week follow-ups, to assess how cannabis exposure modulates immune responses.
Change in serum inflammatory biomarker CRP (pg/mL) | From enrollment to 6 week post-surgery
  The investigators will measure serum biomarker of inflammation CRP (pg/mL) before and after surgery, and again at 2- and 6-week follow-ups, to assess how cannabis exposure modulates immune responses.

SECONDARY OUTCOMES:
Intraoperative opioid dose (MME) | Duration of surgery
  Intraoperative opioid dose (MME) will be extracted from anesthesia records and entered into each patient's individual REDCap record by the study personnel.
Wound healing (cm^2) | From end of surgery to 6 week post-surgery
  Wound healing will be assessed with the aid of the surgical team using the elliptical method, estimating area as (π × length × width)/4 from standardized incision measurements. The investigators will obtain these with the help of the surgical team in the operating room, and then remeasure at follow-up visits.
Postoperative pain scores (0-10) | Post-operative day 0
  Postoperative pain scores will be assessed with the participant using a visual analog scale 0-10, with 0 as no pain and 10 as the greatest amount of pain imaginable. The pain score will be obtained by nurses at 6 hour intervals after surgery till discharge. The data will be extracted from patient health records and entered into their respective records on REDCap.
Mean arterial pressure (MAP) variability minutes | Duration of surgery
  Intraoperative mean arterial pressure (MAP) variability will be measured as the number of minutes the MAP falls under 65 mmHg (i.e., hypotensive) during the surgery. The data will be extracted from patient electronic records and entered into their respective records on REDCap.
Heart rate (HR) variability in minutes | During surgery
  Intraoperative heart rate (HR) variability will be measured as the number of minutes the HR falls under 65 bpm (i.e., bradycardia) or goes above 110 bpm (i.e., tachycardia) during the surgery. The data will be extracted from patient electronic records and entered into their respective records on REDCap.
Total intraoperative vasopressor use (microgram/kg/min) | During surgery
  Intraoperative vasopressor can be administered using multiple different drugs, so the investigators will sum all amounts used into a unified total amount adjusted to micrograms/kg/min. The information will be extracted from anesthesia records and entered into each patient's individual REDCap record by the study personnel.
Postoperative opioid consumption (MME) during hospital stay | Post-operative day 0
  Postoperative opioid consumption (MME) will be extracted patient electronic records and entered into their respective records on REDCap by study personnel.
Pain assessment following discharge | Post-operative day 0 to 6 week post-surgery
  The investigators will use ecological momentary assessments (EMAs) to administered questions remotely in two phases: phase 1 will have EMAs sent once daily for the 1st week following discharge from surgery, and phase 2 will have EMAs sent once weekly between the 2-week and 6-week follow-up sessions. The EMAs will ask patients about pain assessment using the same visual analog scale of 0-10, with 0 as no pain and 10 as the greatest amount of pain imaginable.
Opioid consumption (MME) following discharge | Post-operative day 0 to 6 week post-surgery
  The investigators will use ecological momentary assessments (EMAs) to administered questions remotely in two phases: phase 1 will have EMAs sent once daily for the 1st week following discharge from surgery, and phase 2 will have EMAs sent once weekly between the 2-week and 6-week follow-up sessions. The EMAs will ask patients about medication adherence, patients will be asked to indicate if they took more than their prescribed amount of discharge opiate/analgesic medications and how much (measured in MME).
Cannabis use following discharge | Post-operative day 0 to 6 week post-surgery
  The investigators will use ecological momentary assessments (EMAs) to administered questions remotely in two phases: phase 1 will have EMAs sent once daily for the 1st week following discharge from surgery, and phase 2 will have EMAs sent once weekly between the 2-week and 6-week follow-up sessions. The EMAs will ask participants about if and how much cannabis the participant used (measured in mg) going back 24 hours for phase 1, and 1 week for phase 2.
Cannabis cravings following discharge | Post-operative day 0 to 6 week post-surgery
  The investigators will use ecological momentary assessments (EMAs) to administered questions remotely in two phases: phase 1 will have EMAs sent once daily for the 1st week following discharge from surgery, and phase 2 will have EMAs sent once weekly between the 2-week and 6-week follow-up sessions. The EMAs will ask participants about cannabis cravings with a 4-item Craving Questionnaire going back 24 hours for phase 1, and 1 week for phase 2. The craving questionnaire will ask the participants about intensity, frequency, and length of time of cravings on a scale of 0-4 (0 = None at all; 1= Slight; 2 = Moderate; 3 = Considerable; 4 = Extreme). The fourth question will ask about the total number of times the participants had cravings in the last 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Burger, PhD, Study Director — University of Missouri-Columbia; Randi Foraker, PhD, Study Director — University of Missouri-Columbia
Locations (2):
- United States (2):
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - University Hospital, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No